CLINICAL TRIAL: NCT03760900
Title: Safety of Autologous Cord Blood Cells for Preterm Infants.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, yangjie, Professor, Guangdong Women and Children Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Guang dong WCH
Record Dates: First submitted 2018-11-23; First posted 2018-11-30 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Safety Issues; Effect of Drugs; Neonatal Death
Keywords: Autologous Umbilical Cord Blood Stem Cells; Safety; Effect; neonates; Mechanism
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infusion group (Experimental): Autologous Umbilical Cord Blood Stem Cells Therapy
  Interventions: Combination Product: Autologous Umbilical Cord Blood Stem Cells Therapy

INTERVENTIONS:
Combination Product: Autologous Umbilical Cord Blood Stem Cells Therapy — Autologous Umbilical Cord Blood Stem Cells Therapy,the dose is 5×107cells/kg, within 24 hours after birth

SUMMARY:
To assess the safety of autologous volume- and red blood cell (RBC)-reduced non-cryopreserved umbilical cord blood (UCB) cell infusion to preterm infants.

DETAILED DESCRIPTION:
Preterm birth complications are one of the leading causes of death among children under 5 years of age. Despite advances in medical care, many survivors face a lifetime of disability, including mental and physical retardation, and chronic lung disease. More recently, both allogenic and autogenic cord blood cells have been applied in the treatment of neonatal conditions such as hypoxic-ischemic encephalopathy (HIE) and bronchopulmonary dysplasia (BPD).

Objective-To assess the safety of autologous volume- and red blood cell (RBC)-reduced non-cryopreserved umbilical cord blood (UCB) cell infusion to preterm infants.

Method- This study was a phase I, open-label, single-arm, single center trial to evaluate the safety of autologous, volume- and RBC-reduced non-cyropreserved UCB cell (5×107cells/kg) infusion for preterm infants <37 weeks gestational age. UCB cell characteristics, pre- and post- infusion vital signs, laboratory investigations were recorded. Clinical data including mortality rates and preterm complications were recorded.

Results-After processing, (22.67±4.05) ml UCB cells in volume, (2.67±2.00)×108 cells in number, with (22.67±4.05)×106 CD34+, and (3.72±3.25)×105colony forming cells (CFU-GM), (99.7±0.17%) vitality were infused to 15 preterm infants within 8 hours after birth. No adverse effects were noticed during treatment. All fifteen patients who received UCB infusion survived. The duration of hospitalization ranged from 4 to 65 (30±23.6) days. Regarding preterm complications, no BPD, necrotizing enterocolitis (NEC), retinopathy of prematurity (ROP) were observed. There were 1/15 (7%) infant with intraventricular hemorrhage (IVH), and 5/15 (33.3%) infants with ventilation-associated pneumonia, 10/15(66.67%) with anemia respectively.

Conclusions-Collection, preparation and infusion of fresh autologous UCB cells to preterm infants is feasible and safe. Adequately powered randomized controlled studies are needed.

ELIGIBILITY:
Inborn Infants admitted to the Neonatal Intensive Care Unit (NICU) of Guang Dong Women and Children's Hospital were eligible if they were: 1. Preterm: <37 weeks gestation 2. Without congenital abnormalities; 3. Without maternal chorioamnionitis 4. had available UCB. 5.the mother was negative for hepatitis B (HBsAg and/or HBeAg) and C virus (anti-HCV), syphilis, HIV (anti-HIV-1 and -2) and IgM against cytomegalovirus, rubella, toxoplasma and herpes simplex virus.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2016-06-05 (Actual)

PRIMARY OUTCOMES:
Short-term safety of autologous umbilical cord blood stem cell infusion for preterm infants | during infusion
  1. vital signs
  2. blood gas analysis
  3. blood routine
  4. liver and kidney function before and after infusion will be compared
Short-term safety of autologous umbilical cord blood stem cell infusion for preterm infants | 6 hours after infusion
  1. vital signs
  2. blood gas analysis
  3. blood routine
  4. liver and kidney function before and after infusion will be compared
Long-term safety(2-3 years follow-up after discharge) of autologous umbilical cord blood stem cell infusion for preterm infants | 2years
  1. The growth and development curve will be drawn and compared

CONTACTS AND LOCATIONS:
Overall Officials: jie Yang, PHD, Principal Investigator — Guangdong Women and Children Hospital and Healthy Institutes